CLINICAL TRIAL: NCT01947478
Title: Randomized Trial of MDT-2113 Drug-Eluting Balloon (DEB) vs. Standard PTA for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery and/or Proximal Popliteal Artery
Brief Title: MDT-2113 Drug-Eluting Balloon vs. Standard PTA for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery and/or Proximal Popliteal Artery
Acronym: MDT-2113 SFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10102118DOC
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Femoral Artery Stenosis; Popliteal Artery Stenosis; Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: Drug-Eluting Angioplasty Balloon; Drug Coated Angioplasty Balloon; Peripheral Artery Disease; Experimental; Percutaneous Transluminal Angioplasty (PTA)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDT-2113 Drug-Eluting Balloon (Experimental): Paclitaxel drug-eluting angioplasty balloon
  Interventions: Device: MDT-2113 Drug-Eluting Balloon
- Standard angioplasty balloon (Active Comparator): Standard PTA balloon without Paclitaxel drug-elution
  Interventions: Device: Standard angioplasty balloon

INTERVENTIONS:
Device: MDT-2113 Drug-Eluting Balloon — Subjects will be randomized (2:1) to the MDT-2113 Drug-Eluting Balloon Arm or to the standard non-coated PTA balloon Arm
  Arms: MDT-2113 Drug-Eluting Balloon
Device: Standard angioplasty balloon — Subjects will be randomized (2:1) to the MDT-2113 Drug-Eluting Balloon Arm or to the standard non-coated PTA balloon Arm
  Arms: Standard angioplasty balloon

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of MDT-2113 for the interventional treatment of de novo and non-stented restenotic lesions in the superficial femoral artery (SFA) and the proximal popliteal artery (PPA) as compared to treatment with standard percutaneous transluminal angioplasty (PTA).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 20 years and ≤ 85 years
* Documented ischemia with Rutherford classification 2, 3, or 4
* Able to walk without assistive devices
* Target lesion is in the SFA and/or PPA above the knee
* Target lesion consists of a single de novo or non-stented restenotic lesion (or tandem lesions) or is a combination lesion that meets the following criteria:

  1. ≥ 70% and < 100% occluded with total lesion length ≥ 40 mm and ≤ 200 mm
  2. 100% occluded with total lesion length ≤100 mm
  3. Combination lesions must have total lesion length ≥40 mm and ≤200 mm with an occluded segment that is ≤ 100 mm in length (by visual estimates)
* Reference vessel diameter ≥ 4 mm and ≤7 mm (by visual estimate)
* Angiographic evidence of adequate distal run-off through the foot

Exclusion Criteria:

* Stroke or STEMI within the 3 months prior to enrollment
* Either local or systemic thrombolytic therapy within the 48 hours prior to the index procedure
* Inability to tolerate oral anticoagulation therapy (blood thinners such as warfarin) while on concomitant dual antiplatelet therapy (DAPT)
* Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant/antiplatelet therapies or to paclitaxel, or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure
* Chronic renal insufficiency
* Subject is enrolled in another investigational device, drug, or biologic study
* Any major surgical procedure or intervention performed within the 30-day period prior to or post index procedure
* Contralateral SFA/PPA disease requiring treatment in the same setting as index procedure
* Failure to successfully cross the target lesion
* Angiographic evidence of severe calcification
* Target lesion known in advance of enrollment to require treatment with alternative therapy such as stenting, laser, atherectomy, cryoplasty, brachytherapy, re-entry devices, cutting balloons, scoring balloons; use of embolic protection devices is also prohibited

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Efficacy: Primary patency | 12 month
  Primary patency is defined as freedom from clinically-driven target lesion revascularization (TLR) and freedom from restenosis as determined by duplex ultrasound (DUS)

SECONDARY OUTCOMES:
Primary safety endpoint | 12 month
  Freedom from device- and procedure-related death through 30 days post-procedure, and freedom from target limb major amputation and clinically-driven target vessel revascularization (TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Iida, MD, Principal Investigator — Kansai Rosai Hospital, Amagasaki, Hyogo, Japan
Locations (1):
- Kansai Rosai Hospital, Amagasaki, Hyōgo, Japan

REFERENCES:
- [Derived] Krishnan P, Farhan S, Schneider P, Kamran H, Iida O, Brodmann M, Micari A, Sachar R, Urasawa K, Scheinert D, Ando K, Tarricone A, Doros G, Tepe G, Yokoi H, Laird J, Zeller T. Determinants of Drug-Coated Balloon Failure in Patients Undergoing Femoropopliteal Arterial Intervention. J Am Coll Cardiol. 2022 Sep 27;80(13):1241-1250. doi: 10.1016/j.jacc.2022.06.043. PMID 36137674
- [Derived] Soga Y, Iida O, Urasawa K, Saito S, Jaff MR, Wang H, Ookubo H, Yokoi H. Three-Year Results of the IN.PACT SFA Japan Trial Comparing Drug-Coated Balloons With Percutaneous Transluminal Angioplasty. J Endovasc Ther. 2020 Dec;27(6):946-955. doi: 10.1177/1526602820948240. Epub 2020 Aug 31. PMID 32865145
- [Derived] Shishehbor MH, Schneider PA, Zeller T, Razavi MK, Laird JR, Wang H, Tieche C, Parikh SA, Iida O, Jaff MR. Total IN.PACT drug-coated balloon initiative reporting pooled imaging and propensity-matched cohorts. J Vasc Surg. 2019 Oct;70(4):1177-1191.e9. doi: 10.1016/j.jvs.2019.02.030. PMID 31543165
- [Derived] Schneider PA, Laird JR, Doros G, Gao Q, Ansel G, Brodmann M, Micari A, Shishehbor MH, Tepe G, Zeller T. Mortality Not Correlated With Paclitaxel Exposure: An Independent Patient-Level Meta-Analysis of a Drug-Coated Balloon. J Am Coll Cardiol. 2019 May 28;73(20):2550-2563. doi: 10.1016/j.jacc.2019.01.013. Epub 2019 Jan 25. PMID 30690141
- [Derived] Iida O, Soga Y, Urasawa K, Saito S, Jaff MR, Wang H, Ookubo H, Yokoi H; MDT-2113 SFA Japan Investigators. Drug-Coated Balloon vs Standard Percutaneous Transluminal Angioplasty for the Treatment of Atherosclerotic Lesions in the Superficial Femoral and Proximal Popliteal Arteries: One-Year Results of the MDT-2113 SFA Japan Randomized Trial. J Endovasc Ther. 2018 Feb;25(1):109-117. doi: 10.1177/1526602817745565. Epub 2017 Dec 21. PMID 29264999